CLINICAL TRIAL: NCT04429620
Title: Prospective Assay for SARS-CoV-2 Antibody Detection Indirectly by Immunofluorescence: SARS-CoV2 IIF Method
Brief Title: Prospective Assay for SARS-CoV-2 (COVID-19) Antibody Detection Indirectly by Immunofluorescence: SARS-CoV2 IIF Method
Acronym: IIF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Collaborators: Bilogical Research Centre, Szeged (Unknown)
Responsible Party: Sponsor
Other Study IDs: SARS-CoV-2-IIF-002
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Sars-CoV2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive group: Subjects are diagnosed with SARS-CoV2 by qPCR assay.
  Interventions: Diagnostic Test: Immunfluorescence
- Negative group: Subject were 2 times proved negative SARS-CoV2 by qPCR assay.
  Interventions: Diagnostic Test: Immunfluorescence

INTERVENTIONS:
Diagnostic Test: Immunfluorescence — Serum indirect immunofluorescent (IIF) method is used, analysis is performed under an automated microscope.

SUMMARY:
Prospective assay for SARS-CoV-2 antibody detection indirectly by immunofluorescence: SARS-CoV2 IIF method

DETAILED DESCRIPTION:
Sample preparation, serum separation by centrifugation

* 100 µl of serum for standard SARS-CoV2 ELISA is used according to the instructions for use.
* 100 µl of serum indirect immunofluorescent (IIF) method is used, the samples thus prepared analysis is performed under an automated microscope

ELIGIBILITY:
Inclusion Criteria:

* Person over 18 years of age
* Signing a package leaflet and a informal consent
* In the case of a positive group, confirmed by SARS-CoV2 qPCR Patient with COVID-19 or recovered individual.
* In case of negative group by SARS-CoV2 qPCR test 2 negative in COVID-19 suffering individual

Exclusion Criteria:

* Refuses to sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, Hungarian
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the method by SARS-CoV2 ELISA compared | 8 months
  Sensitivity of the method by SARS-CoV2 ELISA compared

SECONDARY OUTCOMES:
Detectability of the antibodies IgA type against SARS-CoV2 virus | 8 months
  Detectability of the antibodies IgA type against SARS-CoV2 virus in the early stages of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Katalin Burián, MD, Principal Investigator — University of Szeged, Institute of Clinical Microbilogy
Locations (1):
- University of Szeged, Albert Szent-Györgyi Health Center, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: COVID-19 situation update worldwide — https://www.ecdc.europa.eu/en/geographical-distribution-2019-ncov-cases
- See also: COVID-19 CORONAVIRUS PANDEMIC — https://www.worldometers.info/coronavirus/country/italy/
- See also: A serological assay to detect SARS-CoV-2 seroconversion in humans — https://www.medrxiv.org/content/10.1101/2020.03.17.20037713v1.full.pdf
- See also: Serological and molecular findings during SARS-CoV-2 infection: the first case study in Finland, January to February 2020 — https://www.eurosurveillance.org/content/10.2807/1560-7917.ES.2020.25.11.2000266